CLINICAL TRIAL: NCT07014878
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, and Preliminary Efficacy of DCTY1102 Injection in Patients With Advanced Solid Tumors Positive for KRAS G12D Mutation and HLA-A*11:01 Genotype
Brief Title: A Study of DCTY1102 Injection in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing DCTY Biotech Co.,Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2025-009-01
Record Dates: First submitted 2025-05-14; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: PDAC; CRC (Colorectal Cancer); NSCLC; Solid Tumor Malignancies
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Biological: TCR-T therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-T treatment group (Experimental): To evaluate the safety and tolerability of DCTY1102 injection in patients with advanced solid tumors positive for KRAS G12D mutation and genotype HLA-A*11:01, observe potential dose-limiting toxicities (DLTs), determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D), characterize the pharmacokinetic (PK) profile of DCTY1102 injection following infusion, assess its proliferation and persistence in vivo, preliminarily evaluate therapeutic efficacy, and investigate immunogenicity.
  Interventions: Biological: TCR-T cells

INTERVENTIONS:
Biological: TCR-T cells — Dose escalation will follow the standard "3+3" design. Patients will receive a single infusion of DCTY1102 injection. Exploration of higher, lower, or intermediate dose levels may be considered based on emerging safety and tolerability data. Dose escalation will proceed sequentially.

SUMMARY:
This study is an open-label, single-arm, multicenter Phase I clinical trial consisting of a dose-escalation phase (Phase Ia) and a cohort-expansion phase (Phase Ib).

Phase Ia (Dose Escalation) aims to evaluate the safety and tolerability of DCTY1102 Injection in patients with advanced solid tumors positive for KRAS G12D mutation and HLA-A*11:01 genotype, observe potential dose-limiting toxicities (DLTs), determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D), characterize the pharmacokinetic (PK) profile of DCTY1102 following infusion, assess its in vivo proliferation and persistence, preliminarily evaluate therapeutic efficacy, and investigate immunogenicity.

Phase Ib (Cohort Expansion) will be conducted after establishing MTD and/or RP2D in Phase Ia. This phase further evaluates the preliminary efficacy, safety, PK profile, and immunogenicity of DCTY1102 Injection in patients with KRAS G12D mutation-positive, HLA-A*11:01 genotype tumors, including colorectal cancer, pancreatic cancer, or other malignancies. The study plans to establish 2-3 cohorts:

Cohort 1: Colorectal cancer

Cohort 2: Pancreatic cancer

Cohort 3: Other tumor types

Each cohort will enroll approximately 15-31 patients who will receive DCTY1102 infusion at the MTD and/or RP2D dose levels identified in Phase Ia.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent:Written informed consent form (ICF) must be signed prior to any study-related procedures (including pre-screening and main screening).
* Age:18 ≤ Age ≤ 75 years
* Patients with histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors, who have experienced failure of standard treatment (disease progression after treatment or intolerable toxic side effects), have no standard treatment available, for whom standard treatment is not applicable at present, or who refuse standard treatment.
* Have at least one measurable lesion (according to RECIST v1.1).
* The prescreening must meet the following two criteria simultaneously: HLA-A 11:01 genotype, and not carrying the HLA-A 68:01 subtype; Positive for the tumor KRAS G12D mutation.
* ECOG 0-2 with life expectancy ≥3 months.
* LVEF ≥50% by echocardiography
* SpO₂ ≥92% on room air
* Laboratory Parameters: ANC ≥1.5×10⁹/L, ALC ≥0.7×10⁹/L, Platelets ≥75×10⁹/L, Hemoglobin ≥85 g/L, TBIL ≤1.5×ULN, ALT/AST ≤2.5×ULN, Cr ≤1.5×ULN, Ccr ≥50 mL/min, APTT ≤1.5×ULN, INR ≤1.5×ULN
* Child-Pugh Class A or favorable B (score ≤7)
* For patients with advanced primary hepatocellular carcinoma, Child-Pugh liver function classification must be Class A or relatively well-preserved Class B (score ≤7).
* Pre-menopausal fertile women who have not undergone sterilization surgery must agree to use effective contraception from the start of lymphodepleting chemotherapy until one year after cell infusion, and have a negative serum pregnancy test within 14 days before cell infusion
* Men who have not undergone sterilization surgery must agree to use effective contraception from the start of lymphodepleting chemotherapy until one year after cell infusion.

Exclusion Criteria:

* Received last dose of anti - tumor therapy (chemotherapy, endocrine therapy, targeted therapy, immunotherapy, tumor embolization, or traditional Chinese medicine with anti - tumor indications, etc.) within 4 weeks before lymphodepleting chemotherapy.
* Received live - attenuated vaccine within 4 weeks before apheresis.
* Previously received any genetically engineered T - cell therapy or therapy targeting KRAS G12D mutation.
* Known allergy to any component of the study treatment.
* Not recovered from adverse events of previous surgery or therapy to ≤Grade 1 CTCAE v5.0 (excluding any - grade alopecia, ≤Grade 2 peripheral sensory neuropathy, and toxicities deemed safe by the investigator).
* History of leptomeningeal or central nervous system (CNS) metastases, or definite CNS disease within 6 months before cell infusion with residual symptoms. Asymptomatic brain metastases or stable symptoms after treatment (surgery/radiation) without steroid use are allowed.
* Poorly controlled hypertension (systolic BP>160 mmHg and/or diastolic BP>100 mmHg) or clinically significant cardiovascular disease (e.g., stroke, myocardial infarction within 6 months before signing the consent form, unstable angina, NYHA Class Ⅱ or higher heart failure, or severe arrhythmia not controlled by medication or potentially impacting study treatment). ECG shows clinically significant abnormalities in 3 consecutive readings (at least 5 - min intervals) or average QTcF≥450ms.
* Have other severe organic or psychiatric diseases.
* Have systemic active infection requiring IV antibiotics.
* Known HIV infection (anti - HIV antibody - positive), active hepatitis B (HBsAg - positive or HBcAb - positive with HBV - DNA - positive), active hepatitis C (anti - HCV antibody - positive with HCV - RNA - positive), or syphilis infection (anti - TP - positive).
* Diagnosed with severe autoimmune disease requiring long - term (over 2 months) systemic immunosuppressants (steroids) or immune - mediated symptomatic disease (e.g., ulcerative colitis, Crohn's disease, rheumatoid arthritis, SLE, autoimmune vasculitis like Wegener's granulomatosis).
* Used systemic steroids (inhaled or topical use excluded), hydroxyurea, immunomodulators (e.g., α/γ - interferons, GM - CSF, mTOR inhibitors, cyclosporine, thymopeptide, etc.) within 2 weeks before apheresis or plan to use during the study.
* History of allogeneic organ transplantation, allogeneic stem cell transplantation, and renal replacement therapy.
* Uncontrolled diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease, or hepatic failure
* Known alcohol and/or drug abuse.
* Pregnant or breastfeeding women.
* Have any concurrent medical condition or disease that the investigator considers may affect the trial.
* Patients without legal capacity or with limited legal capacity.
* Investigator deems the patient unable to complete all study visits/procedures (including follow - up) or has insufficient adherence, or considers the patient unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of DCTY1102 in subjiects with advanced solid tumors | 28 days after infusion
  Incidence of dose-limiting toxicities
Adverse events and Serious adverse events | up to 24 months post-infusion
  Incidence of adverse events and serious adverse events by dose level

SECONDARY OUTCOMES:
Preliminary anti-tumor activity of DCTY1102 in subject with advanced solid tumors | Up to 24 months post-infusion
  Confirmed ORR per RECIST V1.1,defined as the proportion of subjects with a confirmed PR or better best response

CONTACTS AND LOCATIONS:
Locations (1):
- First Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No